CLINICAL TRIAL: NCT03674177
Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Investigational Unadjuvanted RSV Maternal Vaccine Compared to Placebo When Administered to Healthy Non-pregnant Women.
Brief Title: A Study to Evaluate Different Dose Levels of GlaxoSmithKline (GSK) Biologicals' Investigational Respiratory Syncytial Virus (RSV) Vaccine (GSK3888550A), Based on the Vaccine Safety and the Antibodies (Body Defences) Produced Following Vaccine Administration, When Given to Healthy Non-pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208068; 2018-001340-62 (EudraCT Number)
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Results first posted 2020-04-15 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Vaccines; Safety; Immunogenicity; Reactogenicity; Respiratory Syncytial Viruses
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Observer-blind In this study, the subject and study site personnel involved in the clinical evaluations of the subjects are blinded while other study personnel may be aware of the treatment assignments.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RSV MAT formulation 1 Group (Experimental): Subjects received a single dose (30 µg) injection of the investigational RSV maternal vaccine (GSK3888550A) at Day 1, intramuscularly into the deltoid region of the non-dominant arm
  Interventions: Biological: GSK3888550A RSV Maternal vaccine formulation 1
- RSV MAT formulation 2 Group (Experimental): Subjects received a single dose (60 µg) injection of the investigational RSV maternal vaccine (GSK3888550A) at Day 1, intramuscularly into the deltoid region of the non-dominant arm
  Interventions: Biological: GSK3888550A RSV Maternal vaccine formulation 2
- RSV MAT formulation 3 Group (Experimental): Subjects received a single dose (120 µg) injection of the investigational RSV maternal vaccine (GSK3888550A) at Day 1, intramuscularly into the deltoid region of the non-dominant arm
  Interventions: Biological: GSK3888550A RSV Maternal vaccine formulation 3
- Control Group (Placebo Comparator): Subjects received a single placebo saline injection at Day 1, intramuscularly into the deltoid region of the non-dominant arm
  Interventions: Drug: Placebo (Normal Saline)

INTERVENTIONS:
Biological: GSK3888550A RSV Maternal vaccine formulation 1 — Single dose administered intramuscularly at Day 1 in the deltoid region of the non-dominant arm
  Arms: RSV MAT formulation 1 Group
Biological: GSK3888550A RSV Maternal vaccine formulation 2 — Single dose administered intramuscularly at Day 1 in the deltoid region of the non-dominant arm
  Arms: RSV MAT formulation 2 Group
Biological: GSK3888550A RSV Maternal vaccine formulation 3 — Single dose administered intramuscularly at Day 1 in the deltoid region of the non-dominant arm
  Arms: RSV MAT formulation 3 Group
Drug: Placebo (Normal Saline) — Single dose administered intramuscularly at Day 1 in the deltoid region of the non-dominant arm
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate different dose levels of the investigational RSV maternal vaccine (GSK3888550A) based on safety/reactogenicity and immune response data.

As this is the first time the investigational RSV maternal vaccine (GSK3888550A) is being been used in humans, this study will be performed in healthy non-pregnant women 18-45 years of age before testing in pregnant women.

DETAILED DESCRIPTION:
Healthy non-pregnant women 18-45 years of age will be randomized in a 1:1:1:1 ratio to receive one of three dose levels (30, 60, 120 micrograms [µg]) of the investigational RSV maternal vaccine (GSK3888550A) or placebo, administered as a single intramuscular injection (IM).

There will be a screening visit and five study visits scheduled at Day 1 (study vaccination), Day 8, Day 31, Day 61, and Day 91 to evaluate the primary and secondary objectives of safety/reactogenicity and immunogenicity profiles of the 3 dose levels. Subjects will also be contacted at Day 181. During this contact, the investigator (or delegate) will ask the subject if she has experienced any serious adverse events (SAEs) and or any adverse events (AEs) leading to study withdrawal since the last study visit (Day 360), as well as if she has become pregnant during the post-vaccination period. The investigator (or delegate) will also ask the subject about concomitant vaccinations/products/medications that she has received since the last study visit (D91). Contact should be performed preferably via telephone. Other means of contact (email/other) may be acceptable provided the required information can be fully collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol (e.g. completion of the diary cards/questionnaires, return for follow-up visits, have regular contact to allow evaluation during the study);
* Written informed consent obtained from the subject;
* Healthy female subjects; as established by medical history and clinical examination, aged 18 to 45 years at the time of the vaccination;
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception until 90 days after vaccination

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding vaccination or any planned use during the study period;
* Concurrently participating in the active phase of another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Chronic administration (defined as more than 14 days in total) of immunosuppressant or other immune-modifying drugs, as well as administration of long acting immune modifying drugs, within 6 months prior to the vaccine dose (for corticosteroids, this will mean prednisone higher than or equal to (≥) 5 milligrams per day (mg/day), or equivalent). Inhaled and topical steroids are allowed;
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the study vaccination, or planned administration until 90 days post-vaccination;
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after study vaccination, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before or after study vaccination;
* Previous experimental vaccination against RSV;
* Presence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports;
* Family history of congenital or hereditary immunodeficiency;
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination;
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine;
* Any acute or chronic, clinically significant disease, as determined by physical examination, laboratory screening tests, subject personal report and/or health care provider information. The following conditions will be exclusionary:

  * Diabetes mellitus,
  * Respiratory diseases, such as:

    * Chronic Pulmonary diseases, including Chronic Obstructive Pulmonary Disease (COPD),
    * Bronchopulmonary dysplasia (note: history of past bronchopulmonary dysplasia as a neonate/infant will not be exclusionary),
    * Uncontrolled asthma or asthma necessitating treatment with chronic systemic glucocorticoids
  * Significant and/or uncontrolled psychiatric illness:

    * hospitalization for psychiatric illness, history of suicide attempt(s) or confinement for danger to self or others within 10 years
    * clinically significant depression
  * Major neurological disease including:

    * seizure or adulthood epilepsy (note: history of febrile convulsion in childhood is not exclusionary)
    * myasthenia gravis
    * history of repetitive migraine mal/status migrainosus
  * Significant cardiovascular disease, including:

    * Uncontrolled arterial hypertension,
    * Congenital heart disease (with the exception of corrected atrial or ventricular septal defects),
    * Previous myocardial infarction,
    * Valvular heart disease or history of rheumatic fever,
    * Previous bacterial endocarditis,
    * History of cardiac surgery (with the exception of corrected atrial or ventricular septal defects),
    * Personal or family history of cardiomyopathy or sudden adult death.
  * Known or suspected Hepatitis B or Hepatitis C infection,
  * Any other significant uncontrolled medical illness, defined as any illness requiring new medical and/or surgical treatment or significant modification of treatment dose due to uncontrolled symptoms or drug toxicity, within 3 months prior to study vaccination.
* History of or current autoimmune disease;
* Body mass index (BMI) > 40 Kilograms (kg)/square meters(m^2);
* Pregnant or lactating female;
* Female planning to become pregnant or planning to discontinue contraceptive precautions;
* Hypersensitivity to latex;
* Lymphoproliferative disorder or malignancy within previous 5 years;
* Acute disease and/or fever at the time of enrolment;

  * Fever is defined as temperature ≥ 38°C/100.4°F
  * For subjects with acute disease and/or fever at the time of enrolment, Visit 1 will be rescheduled within the allowed window for the visit.
  * Subjects with fever at screening may be re-screened 1 time at a later date.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Any clinically significant or any ≥ Grade 2* haematological (haemoglobin level, white blood cell, lymphocyte, neutrophil, eosinophil, and platelets) and biochemical (alanine aminotransferase [ALT] aspartate aminotransferase [AST], creatinine, blood urea nitrogen [BUN]) laboratory abnormality detected at the last screening blood sampling; *Grading of laboratory parameters will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials".

For Grade 1 laboratory abnormalities, the investigator should use clinical judgement to decide which ones are clinically relevant.

Subjects with haematological/biochemical values out of normal range at screening which are expected to be temporary, may be re-screened 1 time at a later date.

* Any other condition that the investigator judges may interfere with study procedures or findings;
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe;
* Alcoholism, drug abuse and/or use disorder within the past two years (as defined in Diagnostic and Statistical Manual of Mental Disorders [DSM-5] Diagnostic Criteria);
* Planned move to a location that will prohibit participating in the trial until study end.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The vaccine is for use in pregnant women, as such, the study is female only.
Enrollment: 502 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (2):
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Rochester, New York
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Germany (5):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20864

REFERENCES:
- [Background] Schwarz TF, Johnson C, Grigat C, Apter D, Csonka P, Lindblad N, Nguyen TL, Gao FF, Qian H, Tullio AN, Dieussaert I, Picciolato M, Henry O. Three Dose Levels of a Maternal Respiratory Syncytial Virus Vaccine Candidate Are Well Tolerated and Immunogenic in a Randomized Trial in Nonpregnant Women. J Infect Dis. 2022 Jun 15;225(12):2067-2076. doi: 10.1093/infdis/jiab317. PMID 34146100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 centers in 3 countries: 4 in Finland, 5 in Germany and 2 in the USA.
Pre-assignment Details: Among 579 screened subjects in this study, 77 subjects were screen failure. 502 subjects were enrolled.
Period: Overall Study
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Started | 124 | 126 | 126 | 126
Completed | 122 | 125 | 126 | 124
Not Completed | 2 | 1 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group | Total
Number analyzed (Participants) | 124 | 126 | 126 | 126 | 502
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (7.4) | 32.1 (7.9) | 31.5 (7.6) | 32.2 (7.1) | 32.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 126 | 126 | 126 | 502
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 1 | 1 | 2 | 5 | 9
  BLACK OR AFRICAN AMERICAN | 5 | 5 | 4 | 7 | 21
  OTHER | 3 | 0 | 3 | 0 | 6
  WHITE | 115 | 120 | 117 | 114 | 466

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Adverse Events (AE) During a 7-day Follow-up Period
Description: Assessed solicited local symptoms include pain, redness and swelling, at the injection site. Any = occurrence of the AE regardless of intensity grade. Any Redness and swelling symptom = symptom reported with a surface diameter greater than 20 millimeters.
  Grade 3 pain = significant pain at rest, pain that prevented normal every day activity. Grade 3 redness/swelling = symptom reported with a surface diameter greater than 100 millimeters.
Time Frame: During a 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days)
Population: The analysis was performed on the Exposed Set, which included all subjects with the study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 124 | 125 | 126 | 126
Participants
  Any Pain | 59 | 64 | 67 | 20
  Grade 3 Pain | 1 | 1 | 0 | 0
  Any Redness | 8 | 14 | 10 | 1
  Grade 3 Redness | 0 | 0 | 0 | 0
  Any Swelling | 5 | 7 | 6 | 0
  Grade 3 Swelling | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Adverse Events (AE) During a 7-day Follow-up Period
Description: Assessed solicited general symptoms include fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhea and/or abdominal pain), headache and fever.
  Any Fatigue, gastrointestinal symptoms and headache = occurrence of the symptom regardless of intensity grade and relationship. Any Fever = temperature higher than or equal to 38.0 degrees Celsius (°C), or 100.4 degrees Fahrenheit (°F).
  Grade 3 Fatigue, gastrointestinal symptoms and headache = symptoms that prevented normal activities. Grade 3 Fever = temperature higher than 39.0 degrees Celsius (°C), or 102.2 degrees Fahrenheit (°F).
  Related fatigue, gastrointestinal symptoms, headache and fever(>38°C) = symptoms assessed by the investigator as related to the vaccination.
Time Frame: During a 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 124 | 125 | 126 | 126
Participants
  Any Fatigue | 41 | 49 | 41 | 38
  Grade 3 Fatigue | 3 | 5 | 3 | 4
  Related Fatigue | 25 | 34 | 25 | 27
  Any Gastrointestinal symptoms | 30 | 29 | 23 | 27
  Grade 3 Gastrointestinal symptoms | 2 | 2 | 2 | 1
  Related Gastrointestinal symptoms | 12 | 16 | 13 | 17
  Any Headache | 37 | 51 | 60 | 32
  Grade 3 Headache | 3 | 6 | 2 | 3
  Related Headache | 17 | 25 | 34 | 17
  Any Fever | 2 | 0 | 4 | 0
  Grade 3 Fever | 0 | 0 | 0 | 0
  Related Fever | 0 | 0 | 2 | 0

3. Primary Outcome: Number of Subjects With Any Unsolicited AEs During a 30-day Follow-up Period
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During a 30-day follow-up period after vaccination (i.e., on the day of vaccination and 29 subsequent days)
Population: The analysis was performed on the Exposed Set, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 124 | 126 | 126 | 126
Participants | 45 | 43 | 48 | 44

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) During a 30-day Follow-up Period
Description: Assessed SAEs include any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, or results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 1 (vaccination) up to Day 30 (i.e., on the day of vaccination and 29 subsequent days)
Population: The analysis was performed on the Exposed Set, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 124 | 126 | 126 | 126
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 8
Description: Assessed hematological laboratory parameters include Eosinophils, Hemoglobin, Lymphocytes, Neutrophils, Platelets, White blood cells (WBC). Hematological abnormalities refer to range indicator at timing, categorized as BELOW, WITHIN or ABOVE normal ranges, and compared to baseline range indicator i.e. BELOW(SCR), WITHIN(SCR) or ABOVE(SCR). [e.g. WBC, BELOW(SCR), BELOW = WBC BELOW normal ranges at baseline versus BELOW normal ranges at Day 8].
Time Frame: At Day 8
Population: The analysis was performed on the Exposed Set, which included all vaccinated subjects with available results for the specified laboratory parameter and time point.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 122 | 122 | 125 | 125
Participants
  Eosinophils, BELOW(SCR), BELOW: number analyzed (Participants) | 6 | 5 | 7 | 10
  Eosinophils, BELOW(SCR), BELOW | 2 | 3 | 3 | 8
  Eosinophils, BELOW(SCR), WITHIN: number analyzed (Participants) | 6 | 5 | 7 | 10
  Eosinophils, BELOW(SCR), WITHIN | 4 | 2 | 4 | 2
  Eosinophils, WITHIN(SCR), BELOW: number analyzed (Participants) | 112 | 113 | 117 | 113
  Eosinophils, WITHIN(SCR), BELOW | 3 | 1 | 3 | 3
  Eosinophils, WITHIN(SCR), WITHIN: number analyzed (Participants) | 112 | 113 | 117 | 113
  Eosinophils, WITHIN(SCR), WITHIN | 108 | 109 | 112 | 110
  Eosinophils, WITHIN(SCR), ABOVE: number analyzed (Participants) | 112 | 113 | 117 | 113
  Eosinophils, WITHIN(SCR), ABOVE | 1 | 3 | 2 | 0
  Eosinophils, ABOVE(SCR), WITHIN: number analyzed (Participants) | 4 | 3 | 0 | 2
  Eosinophils, ABOVE(SCR), WITHIN | 2 | 0 | 0 | 1
  Eosinophils, ABOVE(SCR), ABOVE: number analyzed (Participants) | 4 | 3 | 0 | 2
  Eosinophils, ABOVE(SCR), ABOVE | 2 | 3 | 0 | 1
  Hemoglobin, BELOW(SCR), BELOW: number analyzed (Participants) | 7 | 3 | 1 | 2
  Hemoglobin, BELOW(SCR), BELOW | 5 | 2 | 1 | 0
  Hemoglobin, BELOW(SCR), WITHIN: number analyzed (Participants) | 7 | 3 | 1 | 2
  Hemoglobin, BELOW(SCR), WITHIN | 2 | 1 | 0 | 2
  Hemoglobin, WITHIN(SCR), BELOW: number analyzed (Participants) | 115 | 117 | 122 | 122
  Hemoglobin, WITHIN(SCR), BELOW | 2 | 2 | 1 | 5
  Hemoglobin, WITHIN(SCR), WITHIN: number analyzed (Participants) | 115 | 117 | 122 | 122
  Hemoglobin, WITHIN(SCR), WITHIN | 112 | 115 | 120 | 117
  Hemoglobin, WITHIN(SCR), ABOVE: number analyzed (Participants) | 115 | 117 | 122 | 122
  Hemoglobin, WITHIN(SCR), ABOVE | 1 | 0 | 1 | 0
  Hemoglobin, ABOVE(SCR), WITHIN: number analyzed (Participants) | 0 | 2 | 2 | 1
  Hemoglobin, ABOVE(SCR), WITHIN | 0 | 1 | 2 | 0
  Hemoglobin, ABOVE(SCR), ABOVE: number analyzed (Participants) | 0 | 2 | 2 | 1
  Hemoglobin, ABOVE(SCR), ABOVE | 0 | 1 | 0 | 1
  Lymphocytes, BELOW(SCR), WITHIN: number analyzed (Participants) | 0 | 2 | 2 | 0
  Lymphocytes, BELOW(SCR), WITHIN | 0 | 2 | 2 | 0
  Lymphocytes, WITHIN(SCR), BELOW: number analyzed (Participants) | 120 | 118 | 122 | 124
  Lymphocytes, WITHIN(SCR), BELOW | 1 | 1 | 1 | 1
  Lymphocytes, WITHIN(SCR), WITHIN: number analyzed (Participants) | 120 | 118 | 122 | 124
  Lymphocytes, WITHIN(SCR), WITHIN | 119 | 116 | 119 | 121
  Lymphocytes, WITHIN(SCR), ABOVE: number analyzed (Participants) | 120 | 118 | 122 | 124
  Lymphocytes, WITHIN(SCR), ABOVE | 0 | 1 | 2 | 2
  Lymphocytes, ABOVE(SCR), WITHIN: number analyzed (Participants) | 2 | 1 | 0 | 1
  Lymphocytes, ABOVE(SCR), WITHIN | 1 | 0 | 0 | 0
  Lymphocytes, ABOVE(SCR), ABOVE: number analyzed (Participants) | 2 | 1 | 0 | 1
  Lymphocytes, ABOVE(SCR), ABOVE | 1 | 1 | 0 | 1
  Neutrophils, BELOW(SCR), WITHIN: number analyzed (Participants) | 1 | 1 | 0 | 1
  Neutrophils, BELOW(SCR), WITHIN | 1 | 1 | 0 | 1
  Neutrophils, WITHIN(SCR), BELOW: number analyzed (Participants) | 120 | 119 | 120 | 120
  Neutrophils, WITHIN(SCR), BELOW | 2 | 4 | 2 | 1
  Neutrophils, WITHIN(SCR), WITHIN: number analyzed (Participants) | 120 | 119 | 120 | 120
  Neutrophils, WITHIN(SCR), WITHIN | 117 | 111 | 117 | 118
  Neutrophils, WITHIN(SCR), ABOVE: number analyzed (Participants) | 120 | 119 | 120 | 120
  Neutrophils, WITHIN(SCR), ABOVE | 1 | 4 | 1 | 1
  Neutrophils, ABOVE(SCR), WITHIN: number analyzed (Participants) | 1 | 1 | 4 | 4
  Neutrophils, ABOVE(SCR), WITHIN | 1 | 1 | 1 | 3
  Neutrophils, ABOVE(SCR), ABOVE: number analyzed (Participants) | 1 | 1 | 4 | 4
  Neutrophils, ABOVE(SCR), ABOVE | 0 | 0 | 3 | 1
  Platelets, BELOW(SCR), BELOW: number analyzed (Participants) | 0 | 0 | 1 | 2
  Platelets, BELOW(SCR), BELOW | 0 | 0 | 0 | 1
  Platelets, BELOW(SCR), WITHIN: number analyzed (Participants) | 0 | 0 | 1 | 2
  Platelets, BELOW(SCR), WITHIN | 0 | 0 | 1 | 1
  Platelets, WITHIN(SCR), BELOW: number analyzed (Participants) | 118 | 117 | 119 | 116
  Platelets, WITHIN(SCR), BELOW | 1 | 0 | 0 | 0
  Platelets, WITHIN(SCR), WITHIN: number analyzed (Participants) | 118 | 117 | 119 | 116
  Platelets, WITHIN(SCR), WITHIN | 116 | 112 | 115 | 114
  Platelets, WITHIN(SCR), ABOVE: number analyzed (Participants) | 118 | 117 | 119 | 116
  Platelets, WITHIN(SCR), ABOVE | 1 | 5 | 4 | 2
  Platelets, ABOVE(SCR), WITHIN: number analyzed (Participants) | 4 | 5 | 5 | 7
  Platelets, ABOVE(SCR), WITHIN | 3 | 2 | 3 | 3
  Platelets, ABOVE(SCR), ABOVE: number analyzed (Participants) | 4 | 5 | 5 | 7
  Platelets, ABOVE(SCR), ABOVE | 1 | 3 | 2 | 4
  WBC, BELOW(SCR), BELOW: number analyzed (Participants) | 3 | 2 | 5 | 5
  WBC, BELOW(SCR), BELOW | 0 | 1 | 1 | 5
  WBC, BELOW(SCR), WITHIN: number analyzed (Participants) | 3 | 2 | 5 | 5
  WBC, BELOW(SCR), WITHIN | 3 | 1 | 4 | 0
  WBC, WITHIN(SCR), BELOW: number analyzed (Participants) | 118 | 117 | 116 | 115
  WBC, WITHIN(SCR), BELOW | 5 | 4 | 5 | 0
  WBC, WITHIN(SCR), WITHIN: number analyzed (Participants) | 118 | 117 | 116 | 115
  WBC, WITHIN(SCR), WITHIN | 111 | 108 | 108 | 115
  WBC, WITHIN(SCR), ABOVE: number analyzed (Participants) | 118 | 117 | 116 | 115
  WBC, WITHIN(SCR), ABOVE | 2 | 5 | 3 | 0
  WBC, ABOVE(SCR), WITHIN: number analyzed (Participants) | 1 | 3 | 4 | 5
  WBC, ABOVE(SCR), WITHIN | 0 | 1 | 1 | 5
  WBC, ABOVE(SCR), ABOVE: number analyzed (Participants) | 1 | 3 | 4 | 5
  WBC, ABOVE(SCR), ABOVE | 1 | 2 | 3 | 0

6. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 31
Description: Assessed hematological laboratory parameters include Eosinophils, Hemoglobin, Lymphocytes, Neutrophils, Platelets, White blood cells (WBC). Hematological abnormalities refer to range indicator at timing, categorized as BELOW, WITHIN or ABOVE normal ranges, and compared to baseline range indicator i.e. BELOW(SCR), WITHIN(SCR) or ABOVE(SCR) [e.g. WBC, BELOW(SCR), BELOW = WBC BELOW normal ranges at baseline versus BELOW normal ranges at Day 31].
Time Frame: At Day 31
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 121 | 124 | 125 | 125
Participants
  Eosinophils, BELOW(SCR), BELOW: number analyzed (Participants) | 7 | 6 | 8 | 11
  Eosinophils, BELOW(SCR), BELOW | 3 | 3 | 6 | 8
  Eosinophils, BELOW(SCR), WITHIN: number analyzed (Participants) | 7 | 6 | 8 | 11
  Eosinophils, BELOW(SCR), WITHIN | 4 | 3 | 2 | 3
  Eosinophils, WITHIN(SCR), BELOW: number analyzed (Participants) | 110 | 115 | 117 | 112
  Eosinophils, WITHIN(SCR), BELOW | 4 | 2 | 1 | 1
  Eosinophils, WITHIN(SCR), WITHIN: number analyzed (Participants) | 110 | 115 | 117 | 112
  Eosinophils, WITHIN(SCR), WITHIN | 105 | 112 | 115 | 110
  Eosinophils, WITHIN(SCR), ABOVE: number analyzed (Participants) | 110 | 115 | 117 | 112
  Eosinophils, WITHIN(SCR), ABOVE | 1 | 1 | 1 | 1
  Eosinophils, ABOVE(SCR), WITHIN: number analyzed (Participants) | 4 | 3 | 0 | 2
  Eosinophils, ABOVE(SCR), WITHIN | 2 | 1 | 0 | 1
  Eosinophils, ABOVE(SCR), ABOVE: number analyzed (Participants) | 4 | 3 | 0 | 2
  Eosinophils, ABOVE(SCR), ABOVE | 2 | 2 | 0 | 1
  Hemoglobin, BELOW(SCR), BELOW: number analyzed (Participants) | 7 | 3 | 1 | 2
  Hemoglobin, BELOW(SCR), BELOW | 6 | 1 | 1 | 2
  Hemoglobin, BELOW(SCR), WITHIN: number analyzed (Participants) | 7 | 3 | 1 | 2
  Hemoglobin, BELOW(SCR), WITHIN | 1 | 2 | 0 | 0
  Hemoglobin, WITHIN(SCR), BELOW: number analyzed (Participants) | 114 | 118 | 122 | 122
  Hemoglobin, WITHIN(SCR), BELOW | 2 | 4 | 1 | 3
  Hemoglobin, WITHIN(SCR), WITHIN: number analyzed (Participants) | 114 | 118 | 122 | 122
  Hemoglobin, WITHIN(SCR), WITHIN | 112 | 114 | 121 | 119
  Hemoglobin, ABOVE(SCR), WITHIN: number analyzed (Participants) | 0 | 3 | 2 | 1
  Hemoglobin, ABOVE(SCR), WITHIN | 0 | 2 | 1 | 0
  Hemoglobin, ABOVE(SCR), ABOVE: number analyzed (Participants) | 0 | 3 | 2 | 1
  Hemoglobin, ABOVE(SCR), ABOVE | 0 | 1 | 1 | 1
  Lymphocytes, BELOW(SCR), BELOW: number analyzed (Participants) | 0 | 2 | 2 | 0
  Lymphocytes, BELOW(SCR), BELOW | 0 | 1 | 0 | 0
  Lymphocytes, BELOW(SCR), WITHIN: number analyzed (Participants) | 0 | 2 | 2 | 0
  Lymphocytes, BELOW(SCR), WITHIN | 0 | 1 | 2 | 0
  Lymphocytes, WITHIN(SCR), BELOW: number analyzed (Participants) | 119 | 120 | 123 | 124
  Lymphocytes, WITHIN(SCR), BELOW | 0 | 1 | 3 | 2
  Lymphocytes, WITHIN(SCR), WITHIN: number analyzed (Participants) | 119 | 120 | 123 | 124
  Lymphocytes, WITHIN(SCR), WITHIN | 119 | 119 | 119 | 119
  Lymphocytes, WITHIN(SCR), ABOVE: number analyzed (Participants) | 119 | 120 | 123 | 124
  Lymphocytes, WITHIN(SCR), ABOVE | 0 | 0 | 1 | 3
  Lymphocytes, ABOVE(SCR), WITHIN: number analyzed (Participants) | 2 | 2 | 0 | 1
  Lymphocytes, ABOVE(SCR), WITHIN | 2 | 1 | 0 | 0
  Lymphocytes, ABOVE(SCR), ABOVE: number analyzed (Participants) | 2 | 2 | 0 | 1
  Lymphocytes, ABOVE(SCR), ABOVE | 0 | 1 | 0 | 1
  Neutrophils, BELOW(SCR), BELOW: number analyzed (Participants) | 1 | 1 | 0 | 1
  Neutrophils, BELOW(SCR), BELOW | 1 | 0 | 0 | 0
  Neutrophils, BELOW(SCR), WITHIN: number analyzed (Participants) | 1 | 1 | 0 | 1
  Neutrophils, BELOW(SCR), WITHIN | 0 | 1 | 0 | 1
  Neutrophils, WITHIN(SCR), BELOW: number analyzed (Participants) | 119 | 122 | 121 | 120
  Neutrophils, WITHIN(SCR), BELOW | 2 | 2 | 3 | 1
  Neutrophils, WITHIN(SCR), WITHIN: number analyzed (Participants) | 119 | 122 | 121 | 120
  Neutrophils, WITHIN(SCR), WITHIN | 116 | 117 | 114 | 116
  Neutrophils, WITHIN(SCR), ABOVE: number analyzed (Participants) | 119 | 122 | 121 | 120
  Neutrophils, WITHIN(SCR), ABOVE | 1 | 3 | 4 | 3
  Neutrophils, ABOVE(SCR), WITHIN: number analyzed (Participants) | 1 | 1 | 4 | 4
  Neutrophils, ABOVE(SCR), WITHIN | 1 | 0 | 4 | 4
  Neutrophils, ABOVE(SCR), ABOVE: number analyzed (Participants) | 1 | 1 | 4 | 4
  Neutrophils, ABOVE(SCR), ABOVE | 0 | 1 | 0 | 0
  Platelets, BELOW(SCR), BELOW: number analyzed (Participants) | 0 | 0 | 1 | 2
  Platelets, BELOW(SCR), BELOW | 0 | 0 | 0 | 1
  Platelets, BELOW(SCR), WITHIN: number analyzed (Participants) | 0 | 0 | 1 | 2
  Platelets, BELOW(SCR), WITHIN | 0 | 0 | 1 | 1
  Platelets, WITHIN(SCR), BELOW: number analyzed (Participants) | 117 | 119 | 119 | 116
  Platelets, WITHIN(SCR), BELOW | 0 | 0 | 2 | 0
  Platelets, WITHIN(SCR), WITHIN: number analyzed (Participants) | 117 | 119 | 119 | 116
  Platelets, WITHIN(SCR), WITHIN | 115 | 115 | 111 | 113
  Platelets, WITHIN(SCR), ABOVE: number analyzed (Participants) | 117 | 119 | 119 | 116
  Platelets, WITHIN(SCR), ABOVE | 2 | 4 | 6 | 3
  Platelets, ABOVE(SCR), WITHIN: number analyzed (Participants) | 4 | 5 | 5 | 7
  Platelets, ABOVE(SCR), WITHIN | 3 | 1 | 3 | 2
  Platelets, ABOVE(SCR), ABOVE: number analyzed (Participants) | 4 | 5 | 5 | 7
  Platelets, ABOVE(SCR), ABOVE | 1 | 4 | 2 | 5
  WBC, BELOW(SCR), BELOW: number analyzed (Participants) | 3 | 2 | 4 | 5
  WBC, BELOW(SCR), BELOW | 2 | 1 | 2 | 4
  WBC, BELOW(SCR), WITHIN: number analyzed (Participants) | 3 | 2 | 4 | 5
  WBC, BELOW(SCR), WITHIN | 1 | 1 | 2 | 1
  WBC, WITHIN(SCR), BELOW: number analyzed (Participants) | 117 | 119 | 117 | 115
  WBC, WITHIN(SCR), BELOW | 3 | 5 | 9 | 1
  WBC, WITHIN(SCR), WITHIN: number analyzed (Participants) | 117 | 119 | 117 | 115
  WBC, WITHIN(SCR), WITHIN | 109 | 107 | 105 | 110
  WBC, WITHIN(SCR), ABOVE: number analyzed (Participants) | 117 | 119 | 117 | 115
  WBC, WITHIN(SCR), ABOVE | 5 | 7 | 3 | 4
  WBC, ABOVE(SCR), WITHIN: number analyzed (Participants) | 1 | 3 | 4 | 5
  WBC, ABOVE(SCR), WITHIN | 1 | 0 | 4 | 5
  WBC, ABOVE(SCR), ABOVE: number analyzed (Participants) | 1 | 3 | 4 | 5
  WBC, ABOVE(SCR), ABOVE | 0 | 3 | 0 | 0

7. Primary Outcome: Number of Subjects With Biochemical Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 8
Description: Assessed biochemical laboratory parameters include alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN) and creatinine. Biochemical abnormalities refer to range indicator at timing, categorized as BELOW, WITHIN or ABOVE normal ranges, and compared to baseline range indicator i.e. BELOW(SCR), WITHIN(SCR) or ABOVE(SCR)[e.g. ALT, BELOW(SCR), BELOW = ALT BELOW normal ranges at baseline versus BELOW normal ranges at Day 8].
Time Frame: At Day 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 123 | 124 | 126 | 126
Participants
  ALT, BELOW(SCR), WITHIN: number analyzed (Participants) | 0 | 2 | 0 | 0
  ALT, BELOW(SCR), WITHIN | 0 | 2 | 0 | 0
  ALT, WITHIN(SCR), WITHIN: number analyzed (Participants) | 115 | 116 | 123 | 115
  ALT, WITHIN(SCR), WITHIN | 114 | 109 | 120 | 111
  ALT, WITHIN(SCR), ABOVE: number analyzed (Participants) | 115 | 116 | 123 | 115
  ALT, WITHIN(SCR), ABOVE | 1 | 7 | 3 | 4
  ALT, ABOVE(SCR), WITHIN: number analyzed (Participants) | 8 | 6 | 3 | 10
  ALT, ABOVE(SCR), WITHIN | 3 | 6 | 3 | 3
  ALT, ABOVE(SCR), ABOVE: number analyzed (Participants) | 8 | 6 | 3 | 10
  ALT, ABOVE(SCR), ABOVE | 5 | 0 | 0 | 7
  AST, BELOW(SCR), WITHIN: number analyzed (Participants) | 1 | 1 | 2 | 0
  AST, BELOW(SCR), WITHIN | 1 | 1 | 2 | 0
  AST, WITHIN(SCR), BELOW: number analyzed (Participants) | 119 | 122 | 120 | 118
  AST, WITHIN(SCR), BELOW | 0 | 1 | 0 | 0
  AST, WITHIN(SCR), WITHIN: number analyzed (Participants) | 119 | 122 | 120 | 118
  AST, WITHIN(SCR), WITHIN | 116 | 115 | 116 | 116
  AST, WITHIN(SCR), ABOVE: number analyzed (Participants) | 119 | 122 | 120 | 118
  AST, WITHIN(SCR), ABOVE | 3 | 6 | 4 | 2
  AST, ABOVE(SCR), WITHIN: number analyzed (Participants) | 3 | 1 | 4 | 7
  AST, ABOVE(SCR), WITHIN | 3 | 1 | 3 | 6
  AST, ABOVE(SCR), ABOVE: number analyzed (Participants) | 3 | 1 | 4 | 7
  AST, ABOVE(SCR), ABOVE | 0 | 0 | 1 | 1
  BUN, BELOW(SCR), BELOW: number analyzed (Participants) | 4 | 4 | 7 | 1
  BUN, BELOW(SCR), BELOW | 3 | 2 | 3 | 1
  BUN, BELOW(SCR), WITHIN: number analyzed (Participants) | 4 | 4 | 7 | 1
  BUN, BELOW(SCR), WITHIN | 1 | 2 | 4 | 0
  BUN, WITHIN(SCR), BELOW: number analyzed (Participants) | 116 | 119 | 115 | 123
  BUN, WITHIN(SCR), BELOW | 1 | 2 | 2 | 1
  BUN, WITHIN(SCR), WITHIN: number analyzed (Participants) | 116 | 119 | 115 | 123
  BUN, WITHIN(SCR), WITHIN | 113 | 115 | 113 | 121
  BUN, WITHIN(SCR), ABOVE: number analyzed (Participants) | 116 | 119 | 115 | 123
  BUN, WITHIN(SCR), ABOVE | 2 | 2 | 0 | 1
  BUN, ABOVE(SCR), WITHIN: number analyzed (Participants) | 3 | 1 | 3 | 2
  BUN, ABOVE(SCR), WITHIN | 2 | 0 | 3 | 2
  BUN, ABOVE(SCR), ABOVE: number analyzed (Participants) | 3 | 1 | 3 | 2
  BUN, ABOVE(SCR), ABOVE | 1 | 1 | 0 | 0
  Creatinine, BELOW(SCR), BELOW: number analyzed (Participants) | 2 | 3 | 4 | 4
  Creatinine, BELOW(SCR), BELOW | 0 | 1 | 1 | 4
  Creatinine, BELOW(SCR), WITHIN: number analyzed (Participants) | 2 | 3 | 4 | 4
  Creatinine, BELOW(SCR), WITHIN | 2 | 2 | 3 | 0
  Creatinine, WITHIN(SCR), BELOW: number analyzed (Participants) | 119 | 121 | 121 | 121
  Creatinine, WITHIN(SCR), BELOW | 1 | 0 | 1 | 3
  Creatinine, WITHIN(SCR), WITHIN: number analyzed (Participants) | 119 | 121 | 121 | 121
  Creatinine, WITHIN(SCR), WITHIN | 117 | 118 | 119 | 118
  Creatinine, WITHIN(SCR), ABOVE: number analyzed (Participants) | 119 | 121 | 121 | 121
  Creatinine, WITHIN(SCR), ABOVE | 1 | 3 | 1 | 0
  Creatinine, ABOVE(SCR), WITHIN: number analyzed (Participants) | 2 | 0 | 1 | 1
  Creatinine, ABOVE(SCR), WITHIN | 2 | 0 | 1 | 0
  Creatinine, ABOVE(SCR), ABOVE: number analyzed (Participants) | 2 | 0 | 1 | 1
  Creatinine, ABOVE(SCR), ABOVE | 0 | 0 | 0 | 1

8. Primary Outcome: Number of Subjects With Biochemical Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 31
Description: Assessed biochemical laboratory parameters include alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine and blood urea nitrogen (BUN). Biochemical abnormalities refer to range indicator at timing, categorized as BELOW, WITHIN or ABOVE normal ranges, and compared to baseline range indicator i.e. BELOW(SCR), WITHIN(SCR) or ABOVE(SCR) [e.g. ALT, BELOW(SCR), BELOW = ALT BELOW normal ranges at baseline versus BELOW normal ranges at Day 31].
Time Frame: At Day 31
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 123 | 124 | 126 | 126
Participants
  ALT, BELOW(SCR), BELOW: number analyzed (Participants) | 0 | 2 | 0 | 0
  ALT, BELOW(SCR), BELOW | 0 | 1 | 0 | 0
  ALT, BELOW(SCR), WITHIN: number analyzed (Participants) | 0 | 2 | 0 | 0
  ALT, BELOW(SCR), WITHIN | 0 | 1 | 0 | 0
  ALT, WITHIN(SCR), BELOW: number analyzed (Participants) | 115 | 116 | 123 | 116
  ALT, WITHIN(SCR), BELOW | 0 | 0 | 1 | 0
  ALT, WITHIN(SCR), WITHIN: number analyzed (Participants) | 115 | 116 | 123 | 116
  ALT, WITHIN(SCR), WITHIN | 112 | 113 | 121 | 110
  ALT, WITHIN(SCR), ABOVE: number analyzed (Participants) | 115 | 116 | 123 | 116
  ALT, WITHIN(SCR), ABOVE | 3 | 3 | 1 | 6
  ALT, ABOVE(SCR), WITHIN: number analyzed (Participants) | 8 | 6 | 3 | 10
  ALT, ABOVE(SCR), WITHIN | 4 | 5 | 3 | 6
  ALT, ABOVE(SCR), ABOVE: number analyzed (Participants) | 8 | 6 | 3 | 10
  ALT, ABOVE(SCR), ABOVE | 4 | 1 | 0 | 4
  AST, BELOW(SCR), WITHIN: number analyzed (Participants) | 1 | 1 | 2 | 0
  AST, BELOW(SCR), WITHIN | 1 | 1 | 2 | 0
  AST, WITHIN(SCR), BELOW: number analyzed (Participants) | 119 | 122 | 120 | 119
  AST, WITHIN(SCR), BELOW | 0 | 0 | 0 | 1
  AST, WITHIN(SCR), WITHIN: number analyzed (Participants) | 119 | 122 | 120 | 119
  AST, WITHIN(SCR), WITHIN | 115 | 118 | 120 | 114
  AST, WITHIN(SCR), ABOVE: number analyzed (Participants) | 119 | 122 | 120 | 119
  AST, WITHIN(SCR), ABOVE | 4 | 4 | 0 | 4
  AST, ABOVE(SCR), WITHIN: number analyzed (Participants) | 3 | 1 | 4 | 7
  AST, ABOVE(SCR), WITHIN | 3 | 1 | 3 | 6
  AST, ABOVE(SCR), ABOVE: number analyzed (Participants) | 3 | 1 | 4 | 7
  AST, ABOVE(SCR), ABOVE | 0 | 0 | 1 | 1
  BUN, BELOW(SCR), BELOW: number analyzed (Participants) | 4 | 4 | 7 | 1
  BUN, BELOW(SCR), BELOW | 2 | 2 | 2 | 1
  BUN, BELOW(SCR), WITHIN: number analyzed (Participants) | 4 | 4 | 7 | 1
  BUN, BELOW(SCR), WITHIN | 2 | 2 | 5 | 0
  BUN, WITHIN(SCR), BELOW: number analyzed (Participants) | 116 | 119 | 116 | 123
  BUN, WITHIN(SCR), BELOW | 2 | 2 | 0 | 2
  BUN, WITHIN(SCR), WITHIN: number analyzed (Participants) | 116 | 119 | 116 | 123
  BUN, WITHIN(SCR), WITHIN | 113 | 117 | 115 | 120
  BUN, WITHIN(SCR), ABOVE: number analyzed (Participants) | 116 | 119 | 116 | 123
  BUN, WITHIN(SCR), ABOVE | 1 | 0 | 1 | 1
  BUN, ABOVE(SCR), WITHIN: number analyzed (Participants) | 3 | 1 | 3 | 2
  BUN, ABOVE(SCR), WITHIN | 3 | 0 | 3 | 2
  BUN, ABOVE(SCR), ABOVE: number analyzed (Participants) | 3 | 1 | 3 | 2
  BUN, ABOVE(SCR), ABOVE | 0 | 1 | 0 | 0
  Creatinine, BELOW(SCR), BELOW: number analyzed (Participants) | 2 | 3 | 4 | 4
  Creatinine, BELOW(SCR), BELOW | 0 | 0 | 0 | 3
  Creatinine, BELOW(SCR), WITHIN: number analyzed (Participants) | 2 | 3 | 4 | 4
  Creatinine, BELOW(SCR), WITHIN | 2 | 3 | 4 | 1
  Creatinine, WITHIN(SCR), BELOW: number analyzed (Participants) | 119 | 121 | 121 | 121
  Creatinine, WITHIN(SCR), BELOW | 0 | 1 | 0 | 2
  Creatinine, WITHIN(SCR), WITHIN: number analyzed (Participants) | 119 | 121 | 121 | 121
  Creatinine, WITHIN(SCR), WITHIN | 118 | 116 | 117 | 116
  Creatinine, WITHIN(SCR), ABOVE: number analyzed (Participants) | 119 | 121 | 121 | 121
  Creatinine, WITHIN(SCR), ABOVE | 1 | 4 | 4 | 3
  Creatinine, ABOVE(SCR), WITHIN: number analyzed (Participants) | 2 | 0 | 1 | 1
  Creatinine, ABOVE(SCR), WITHIN | 1 | 0 | 1 | 0
  Creatinine, ABOVE(SCR), ABOVE: number analyzed (Participants) | 2 | 0 | 1 | 1
  Creatinine, ABOVE(SCR), ABOVE | 1 | 0 | 0 | 1

9. Primary Outcome: Number of Subjects With Hematological Laboratory Results Versus Baseline, by Maximum Grading, at Day 8
Description: Assessed hematological laboratory parameters include Eosinophils, Hemoglobin, Lymphocytes Decrease, Neutrophils Decrease, Platelets Decrease, WBC Decrease and WBC Increase, as graded by the Food and Drug Administration [FDA] Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Assessed grades at specified time point, are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = life threatening, as compared to the baseline status of the same parameter, at baseline [e.g. WBC decrease-Grade 1(SCR)-Grade 1 = WBC decrease Grade 1 at baseline versus Grade 1 at Day 8]. "Any" corresponding to any grade and "Grade 0" to normal ranges.
Time Frame: At Day 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 122 | 122 | 125 | 125
Participants
  Eosinophils, Any(SCR), GRADE 0: number analyzed (Participants) | 122 | 121 | 124 | 125
  Eosinophils, Any(SCR), GRADE 0 | 121 | 120 | 124 | 125
  Eosinophils, Any(SCR), GRADE 1: number analyzed (Participants) | 122 | 121 | 124 | 125
  Eosinophils, Any(SCR), GRADE 1 | 1 | 0 | 0 | 0
  Eosinophils, Any(SCR), GRADE 2: number analyzed (Participants) | 122 | 121 | 124 | 125
  Eosinophils, Any(SCR), GRADE 2 | 0 | 1 | 0 | 0
  Eosinophils, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 120 | 120 | 124 | 123
  Eosinophils, Grade 0(SCR), GRADE 0 | 119 | 120 | 124 | 123
  Eosinophils, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 120 | 120 | 124 | 123
  Eosinophils, Grade 0(SCR), GRADE 1 | 1 | 0 | 0 | 0
  Eosinophils, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 2 | 1 | 0 | 2
  Eosinophils, Grade 1(SCR), GRADE 0 | 2 | 0 | 0 | 2
  Eosinophils, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 2 | 1 | 0 | 2
  Eosinophils, Grade 1(SCR), GRADE 2 | 0 | 1 | 0 | 0
  Hemoglobin, Any(SCR), GRADE 0 | 110 | 111 | 114 | 110
  Hemoglobin, Any(SCR), GRADE 1 | 11 | 9 | 10 | 15
  Hemoglobin, Any(SCR), GRADE 2 | 1 | 2 | 1 | 0
  Hemoglobin, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 110 | 111 | 115 | 116
  Hemoglobin, Grade 0(SCR), GRADE 0 | 106 | 107 | 110 | 106
  Hemoglobin, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 110 | 111 | 115 | 116
  Hemoglobin, Grade 0(SCR), GRADE 1 | 4 | 4 | 5 | 10
  Hemoglobin, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 11 | 11 | 10 | 9
  Hemoglobin, Grade 1(SCR), GRADE 0 | 4 | 4 | 4 | 4
  Hemoglobin, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 11 | 11 | 10 | 9
  Hemoglobin, Grade 1(SCR), GRADE 1 | 7 | 5 | 5 | 5
  Hemoglobin, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 11 | 11 | 10 | 9
  Hemoglobin, Grade 1(SCR), GRADE 2 | 0 | 2 | 1 | 0
  Hemoglobin, Grade 2(SCR), GRADE 2: number analyzed (Participants) | 1 | 0 | 0 | 0
  Hemoglobin, Grade 2(SCR), GRADE 2 | 1 | 0 | 0 | 0
  Lymphocytes Decrease, Any(SCR), GRADE 0: number analyzed (Participants) | 122 | 121 | 124 | 125
  Lymphocytes Decrease, Any(SCR), GRADE 0 | 120 | 118 | 122 | 122
  Lymphocytes Decrease, Any(SCR), GRADE 1: number analyzed (Participants) | 122 | 121 | 124 | 125
  Lymphocytes Decrease, Any(SCR), GRADE 1 | 1 | 2 | 2 | 3
  Lymphocytes Decrease, Any(SCR), GRADE 2: number analyzed (Participants) | 122 | 121 | 124 | 125
  Lymphocytes Decrease, Any(SCR), GRADE 2 | 1 | 1 | 0 | 0
  Lymphocytes Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 122 | 119 | 120 | 120
  Lymphocytes Decrease, Grade 0(SCR), GRADE 0 | 120 | 117 | 118 | 120
  Lymphocytes Decrease, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 122 | 119 | 120 | 120
  Lymphocytes Decrease, Grade 0(SCR), GRADE 1 | 1 | 1 | 2 | 0
  Lymphocytes Decrease, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 122 | 119 | 120 | 120
  Lymphocytes Decrease, Grade 0(SCR), GRADE 2 | 1 | 1 | 0 | 0
  Lymphocytes Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 0 | 2 | 3 | 5
  Lymphocytes Decrease, Grade 1(SCR), GRADE 0 | 0 | 1 | 3 | 2
  Lymphocytes Decrease, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 0 | 2 | 3 | 5
  Lymphocytes Decrease, Grade 1(SCR), GRADE 1 | 0 | 1 | 0 | 3
  Lymphocytes Decrease, Grade 2(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes Decrease, Grade 2(SCR), GRADE 0 | 0 | 0 | 1 | 0
  Neutrophils Decrease, Any(SCR), GRADE 0: number analyzed (Participants) | 122 | 121 | 124 | 125
  Neutrophils Decrease, Any(SCR), GRADE 0 | 112 | 113 | 116 | 118
  Neutrophils Decrease, Any(SCR), GRADE 1: number analyzed (Participants) | 122 | 121 | 124 | 125
  Neutrophils Decrease, Any(SCR), GRADE 1 | 10 | 5 | 8 | 6
  Neutrophils Decrease, Any(SCR), GRADE 2: number analyzed (Participants) | 122 | 121 | 124 | 125
  Neutrophils Decrease, Any(SCR), GRADE 2 | 0 | 3 | 0 | 1
  Neutrophils Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 117 | 115 | 119 | 119
  Neutrophils Decrease, Grade 0(SCR), GRADE 0 | 109 | 109 | 111 | 115
  Neutrophils Decrease, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 117 | 115 | 119 | 119
  Neutrophils Decrease, Grade 0(SCR), GRADE 1 | 8 | 4 | 8 | 4
  Neutrophils Decrease, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 117 | 115 | 119 | 119
  Neutrophils Decrease, Grade 0(SCR), GRADE 2 | 0 | 2 | 0 | 0
  Neutrophils Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 4 | 6 | 5 | 6
  Neutrophils Decrease, Grade 1(SCR), GRADE 0 | 3 | 4 | 5 | 3
  Neutrophils Decrease, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 4 | 6 | 5 | 6
  Neutrophils Decrease, Grade 1(SCR), GRADE 1 | 1 | 1 | 0 | 2
  Neutrophils Decrease, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 4 | 6 | 5 | 6
  Neutrophils Decrease, Grade 1(SCR), GRADE 2 | 0 | 1 | 0 | 1
  Neutrophils Decrease, Grade 2(SCR), GRADE 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Neutrophils Decrease, Grade 2(SCR), GRADE 1 | 1 | 0 | 0 | 0
  Platelets Decrease, Any(SCR), GRADE 0 | 121 | 122 | 125 | 125
  Platelets Decrease, Any(SCR), GRADE 1 | 1 | 0 | 0 | 0
  Platelets Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 122 | 122 | 125 | 123
  Platelets Decrease, Grade 0(SCR), GRADE 0 | 121 | 122 | 125 | 123
  Platelets Decrease, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 122 | 122 | 125 | 123
  Platelets Decrease, Grade 0(SCR), GRADE 1 | 1 | 0 | 0 | 0
  Platelets Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 2
  Platelets Decrease, Grade 1(SCR), GRADE 0 | 0 | 0 | 0 | 2
  WBC Decrease, Any(SCR), GRADE 0 | 121 | 119 | 125 | 124
  WBC Decrease, Any(SCR), GRADE 1 | 1 | 3 | 0 | 1
  WBC Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 121 | 121 | 124 | 121
  WBC Decrease, Grade 0(SCR), GRADE 0 | 120 | 118 | 124 | 120
  WBC Decrease, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 121 | 121 | 124 | 121
  WBC Decrease, Grade 0(SCR), GRADE 1 | 1 | 3 | 0 | 1
  WBC Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 1 | 1 | 1 | 4
  WBC Decrease, Grade 1(SCR), GRADE 0 | 1 | 1 | 1 | 4
  WBC Increase, Any(SCR), GRADE 0 | 119 | 118 | 121 | 125
  WBC Increase, Any(SCR), GRADE 1 | 3 | 3 | 4 | 0
  WBC Increase, Any(SCR), GRADE 2 | 0 | 1 | 0 | 0
  WBC Increase, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 119 | 118 | 121 | 122
  WBC Increase, Grade 0(SCR), GRADE 0 | 118 | 116 | 120 | 122
  WBC Increase, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 119 | 118 | 121 | 122
  WBC Increase, Grade 0(SCR), GRADE 1 | 1 | 2 | 1 | 0
  WBC Increase, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 3 | 4 | 4 | 3
  WBC Increase, Grade 1(SCR), GRADE 0 | 1 | 2 | 1 | 3
  WBC Increase, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 3 | 4 | 4 | 3
  WBC Increase, Grade 1(SCR), GRADE 1 | 2 | 1 | 3 | 0
  WBC Increase, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 3 | 4 | 4 | 3
  WBC Increase, Grade 1(SCR), GRADE 2 | 0 | 1 | 0 | 0

10. Primary Outcome: Number of Subjects With Hematological Laboratory Results Versus Baseline, by Maximum Grading, at Day 31
Description: Assessed hematological laboratory parameters include Eosinophils, Hemoglobin, Lymphocytes Decrease, Neutrophils Decrease, Platelets Decrease, WBC Decrease and WBC Increase, as graded by the Food and Drug Administration [FDA] Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Assessed grades at specified time point, are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = life threatening, as compared to the baseline status of the same parameter, at baseline [e.g. WBC decrease-Grade 1(SCR)-Grade 1 = WBC decrease Grade 1 at baseline versus Grade 1 at Day 31]. "Any" corresponding to any grade and "Grade 0" to normal ranges.
Time Frame: At Day 31
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 121 | 124 | 125 | 125
Participants
  Eosinophils, Any(SCR), GRADE 0 | 118 | 122 | 125 | 125
  Eosinophils, Any(SCR), GRADE 1 | 3 | 2 | 0 | 0
  Eosinophils, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 119 | 123 | 125 | 123
  Eosinophils, Grade 0(SCR), GRADE 0 | 117 | 122 | 125 | 123
  Eosinophils, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 119 | 123 | 125 | 123
  Eosinophils, Grade 0(SCR), GRADE 1 | 2 | 1 | 0 | 0
  Eosinophils, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 2 | 1 | 0 | 2
  Eosinophils, Grade 1(SCR), GRADE 0 | 1 | 0 | 0 | 2
  Eosinophils, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 2 | 1 | 0 | 2
  Eosinophils, Grade 1(SCR), GRADE 1 | 1 | 1 | 0 | 0
  Hemoglobin, Any(SCR), GRADE 0 | 108 | 115 | 112 | 114
  Hemoglobin, Any(SCR), GRADE 1 | 11 | 7 | 13 | 8
  Hemoglobin, Any(SCR), GRADE 2 | 2 | 2 | 0 | 3
  Hemoglobin, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 110 | 113 | 115 | 116
  Hemoglobin, Grade 0(SCR), GRADE 0 | 106 | 112 | 109 | 111
  Hemoglobin, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 110 | 113 | 115 | 116
  Hemoglobin, Grade 0(SCR), GRADE 1 | 4 | 1 | 6 | 3
  Hemoglobin, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 110 | 113 | 115 | 116
  Hemoglobin, Grade 0(SCR), GRADE 2 | 0 | 0 | 0 | 2
  Hemoglobin, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 10 | 11 | 10 | 9
  Hemoglobin, Grade 1(SCR), GRADE 0 | 2 | 3 | 3 | 3
  Hemoglobin, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 10 | 11 | 10 | 9
  Hemoglobin, Grade 1(SCR), GRADE 1 | 7 | 6 | 7 | 5
  Hemoglobin, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 10 | 11 | 10 | 9
  Hemoglobin, Grade 1(SCR), GRADE 2 | 1 | 2 | 0 | 1
  Hemoglobin, Grade 2(SCR), GRADE 2: number analyzed (Participants) | 1 | 0 | 0 | 0
  Hemoglobin, Grade 2(SCR), GRADE 2 | 1 | 0 | 0 | 0
  Lymphocytes Decrease, Any(SCR), GRADE 0 | 119 | 119 | 121 | 120
  Lymphocytes Decrease, Any(SCR), GRADE 1 | 2 | 5 | 4 | 4
  Lymphocytes Decrease, Any(SCR), GRADE 2 | 0 | 0 | 0 | 1
  Lymphocytes Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 121 | 122 | 121 | 120
  Lymphocytes Decrease, Grade 0(SCR), GRADE 0 | 119 | 118 | 117 | 117
  Lymphocytes Decrease, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 121 | 122 | 121 | 120
  Lymphocytes Decrease, Grade 0(SCR), GRADE 1 | 2 | 4 | 4 | 3
  Lymphocytes Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 0 | 2 | 3 | 5
  Lymphocytes Decrease, Grade 1(SCR), GRADE 0 | 0 | 1 | 3 | 3
  Lymphocytes Decrease, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 0 | 2 | 3 | 5
  Lymphocytes Decrease, Grade 1(SCR), GRADE 1 | 0 | 1 | 0 | 1
  Lymphocytes Decrease, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 0 | 2 | 3 | 5
  Lymphocytes Decrease, Grade 1(SCR), GRADE 2 | 0 | 0 | 0 | 1
  Lymphocytes Decrease, Grade 2(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes Decrease, Grade 2(SCR), GRADE 0 | 0 | 0 | 1 | 0
  Neutrophils Decrease, Any(SCR), GRADE 0 | 111 | 115 | 114 | 116
  Neutrophils Decrease, Any(SCR), GRADE 1 | 8 | 7 | 10 | 8
  Neutrophils Decrease, Any(SCR), GRADE 2 | 1 | 2 | 1 | 1
  Neutrophils Decrease, Any(SCR), GRADE 3 | 1 | 0 | 0 | 0
  Neutrophils Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 117 | 118 | 120 | 119
  Neutrophils Decrease, Grade 0(SCR), GRADE 0 | 109 | 112 | 109 | 114
  Neutrophils Decrease, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 117 | 118 | 120 | 119
  Neutrophils Decrease, Grade 0(SCR), GRADE 1 | 7 | 5 | 10 | 4
  Neutrophils Decrease, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 117 | 118 | 120 | 119
  Neutrophils Decrease, Grade 0(SCR), GRADE 2 | 0 | 1 | 1 | 1
  Neutrophils Decrease, Grade 0(SCR), GRADE 3: number analyzed (Participants) | 117 | 118 | 120 | 119
  Neutrophils Decrease, Grade 0(SCR), GRADE 3 | 1 | 0 | 0 | 0
  Neutrophils Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 3 | 6 | 5 | 6
  Neutrophils Decrease, Grade 1(SCR), GRADE 0 | 2 | 3 | 5 | 2
  Neutrophils Decrease, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 3 | 6 | 5 | 6
  Neutrophils Decrease, Grade 1(SCR), GRADE 1 | 1 | 2 | 0 | 4
  Neutrophils Decrease, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 3 | 6 | 5 | 6
  Neutrophils Decrease, Grade 1(SCR), GRADE 2 | 0 | 1 | 0 | 0
  Neutrophils Decrease, Grade 2(SCR), GRADE 2: number analyzed (Participants) | 1 | 0 | 0 | 0
  Neutrophils Decrease, Grade 2(SCR), GRADE 2 | 1 | 0 | 0 | 0
  Platelets Decrease, Any(SCR), GRADE 0 | 121 | 124 | 125 | 125
  Platelets Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 121 | 124 | 125 | 123
  Platelets Decrease, Grade 0(SCR), GRADE 0 | 121 | 124 | 125 | 123
  Platelets Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 2
  Platelets Decrease, Grade 1(SCR), GRADE 0 | 0 | 0 | 0 | 2
  WBC Decrease, Any(SCR), GRADE 0 | 119 | 122 | 121 | 123
  WBC Decrease, Any(SCR), GRADE 1 | 2 | 2 | 4 | 2
  WBC Decrease, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 120 | 123 | 124 | 121
  WBC Decrease, Grade 0(SCR), GRADE 0 | 119 | 121 | 120 | 120
  WBC Decrease, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 120 | 123 | 124 | 121
  WBC Decrease, Grade 0(SCR), GRADE 1 | 1 | 2 | 4 | 1
  WBC Decrease, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 1 | 1 | 1 | 4
  WBC Decrease, Grade 1(SCR), GRADE 0 | 0 | 1 | 1 | 3
  WBC Decrease, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 1 | 1 | 1 | 4
  WBC Decrease, Grade 1(SCR), GRADE 1 | 1 | 0 | 0 | 1
  WBC Increase, Any(SCR), GRADE 0 | 120 | 116 | 122 | 122
  WBC Increase, Any(SCR), GRADE 1 | 1 | 8 | 3 | 3
  WBC Increase, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 118 | 120 | 121 | 122
  WBC Increase, Grade 0(SCR), GRADE 0 | 118 | 115 | 118 | 119
  WBC Increase, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 118 | 120 | 121 | 122
  WBC Increase, Grade 0(SCR), GRADE 1 | 0 | 5 | 3 | 3
  WBC Increase, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 3 | 4 | 4 | 3
  WBC Increase, Grade 1(SCR), GRADE 0 | 2 | 1 | 4 | 3
  WBC Increase, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 3 | 4 | 4 | 3
  WBC Increase, Grade 1(SCR), GRADE 1 | 1 | 3 | 0 | 0

11. Primary Outcome: Number of Subjects With Biochemical Laboratory Results Versus Baseline, by Maximum Grading, at Day 8
Description: Assessed biochemical laboratory parameters include alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN) and creatinine, as graded by the Food and Drug Administration [FDA] Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Assessed grades at specified time point, are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = life threatening, as compared to the baseline status of the same parameter, at baseline [e.g. ALT-Grade 1(SCR)-Grade 1 = ALT Grade 1 at baseline versus Grade 1 at Day 8]. "Any" corresponding to any grade and "Grade 0" to normal ranges.
Time Frame: At Day 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 123 | 124 | 126 | 126
Participants
  ALT - increase by factor, Any(SCR), GRADE 0: number analyzed (Participants) | 123 | 124 | 126 | 125
  ALT - increase by factor, Any(SCR), GRADE 0 | 118 | 119 | 124 | 117
  ALT - increase by factor, Any(SCR), GRADE 1: number analyzed (Participants) | 123 | 124 | 126 | 125
  ALT - increase by factor, Any(SCR), GRADE 1 | 5 | 3 | 1 | 7
  ALT - increase by factor, Any(SCR), GRADE 2: number analyzed (Participants) | 123 | 124 | 126 | 125
  ALT - increase by factor, Any(SCR), GRADE 2 | 0 | 1 | 1 | 0
  ALT - increase by factor, Any(SCR), GRADE 3: number analyzed (Participants) | 123 | 124 | 126 | 125
  ALT - increase by factor, Any(SCR), GRADE 3 | 0 | 1 | 0 | 1
  ALT - increase by factor, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 116 | 120 | 123 | 116
  ALT - increase by factor, Grade 0(SCR), GRADE 0 | 115 | 115 | 121 | 114
  ALT - increase by factor, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 116 | 120 | 123 | 116
  ALT - increase by factor, Grade 0(SCR), GRADE 1 | 1 | 3 | 1 | 2
  ALT - increase by factor, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 116 | 120 | 123 | 116
  ALT - increase by factor, Grade 0(SCR), GRADE 2 | 0 | 1 | 1 | 0
  ALT - increase by factor, Grade 0(SCR), GRADE 3: number analyzed (Participants) | 116 | 120 | 123 | 116
  ALT - increase by factor, Grade 0(SCR), GRADE 3 | 0 | 1 | 0 | 0
  ALT - increase by factor, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 6 | 4 | 3 | 9
  ALT - increase by factor, Grade 1(SCR), GRADE 0 | 3 | 4 | 3 | 3
  ALT - increase by factor, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 6 | 4 | 3 | 9
  ALT - increase by factor, Grade 1(SCR), GRADE 1 | 3 | 0 | 0 | 5
  ALT - increase by factor, Grade 1(SCR), GRADE 3: number analyzed (Participants) | 6 | 4 | 3 | 9
  ALT - increase by factor, Grade 1(SCR), GRADE 3 | 0 | 0 | 0 | 1
  ALT - increase by factor, Grade 2(SCR), GRADE 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  ALT - increase by factor, Grade 2(SCR), GRADE 1 | 1 | 0 | 0 | 0
  AST - increase by factor, Any(SCR), GRADE 0: number analyzed (Participants) | 123 | 124 | 126 | 125
  AST - increase by factor, Any(SCR), GRADE 0 | 123 | 120 | 124 | 122
  AST - increase by factor, Any(SCR), GRADE 1: number analyzed (Participants) | 123 | 124 | 126 | 125
  AST - increase by factor, Any(SCR), GRADE 1 | 0 | 3 | 2 | 3
  AST - increase by factor, Any(SCR), GRADE 3: number analyzed (Participants) | 123 | 124 | 126 | 125
  AST - increase by factor, Any(SCR), GRADE 3 | 0 | 1 | 0 | 0
  AST - increase by factor, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 120 | 123 | 125 | 121
  AST - increase by factor, Grade 0(SCR), GRADE 0 | 120 | 119 | 124 | 119
  AST - increase by factor, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 120 | 123 | 125 | 121
  AST - increase by factor, Grade 0(SCR), GRADE 1 | 0 | 3 | 1 | 2
  AST - increase by factor, Grade 0(SCR), GRADE 3: number analyzed (Participants) | 120 | 123 | 125 | 121
  AST - increase by factor, Grade 0(SCR), GRADE 3 | 0 | 1 | 0 | 0
  AST - increase by factor, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 3 | 1 | 1 | 4
  AST - increase by factor, Grade 1(SCR), GRADE 0 | 3 | 1 | 0 | 3
  AST - increase by factor, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 3 | 1 | 1 | 4
  AST - increase by factor, Grade 1(SCR), GRADE 1 | 0 | 0 | 1 | 1
  Blood Urea Nitrogen, Any(SCR), GRADE 0: number analyzed (Participants) | 123 | 124 | 125 | 126
  Blood Urea Nitrogen, Any(SCR), GRADE 0 | 122 | 123 | 124 | 125
  Blood Urea Nitrogen, Any(SCR), GRADE 1: number analyzed (Participants) | 123 | 124 | 125 | 126
  Blood Urea Nitrogen, Any(SCR), GRADE 1 | 1 | 1 | 1 | 0
  Blood Urea Nitrogen, Any(SCR), GRADE 2: number analyzed (Participants) | 123 | 124 | 125 | 126
  Blood Urea Nitrogen, Any(SCR), GRADE 2 | 0 | 0 | 0 | 1
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 123 | 124 | 124 | 125
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 0 | 122 | 123 | 123 | 124
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 123 | 124 | 124 | 125
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 1 | 1 | 1 | 1 | 0
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 123 | 124 | 124 | 125
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 2 | 0 | 0 | 0 | 1
  Blood Urea Nitrogen, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Blood Urea Nitrogen, Grade 1(SCR), GRADE 0 | 0 | 0 | 1 | 0
  Blood Urea Nitrogen, Grade 2(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 1
  Blood Urea Nitrogen, Grade 2(SCR), GRADE 0 | 0 | 0 | 0 | 1
  Creatinine, Any(SCR), GRADE 0 | 122 | 124 | 126 | 126
  Creatinine, Any(SCR), GRADE 3 | 1 | 0 | 0 | 0
  Creatinine, Grade 0(SCR), GRADE 0 | 122 | 124 | 126 | 126
  Creatinine, Grade 0(SCR), GRADE 3 | 1 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects With Biochemical Laboratory Results Versus Baseline, by Maximum Grading, at Day 31
Description: Assessed biochemical laboratory parameters include alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN) and creatinine, as graded by the Food and Drug Administration [FDA] Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Assessed grades at specified time point, are Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe and Grade 4 = life threatening, as compared to the baseline status of the same parameter, at baseline [e.g. ALT-Grade 1(SCR)-Grade 1 = ALT Grade 1 at baseline versus Grade 1 at Day 31]. "Any" corresponding to any grade and "Grade 0" to normal ranges.
Time Frame: At Day 31
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 123 | 124 | 126 | 126
Participants
  ALT - increase by factor, Any(SCR), GRADE 0 | 117 | 121 | 125 | 118
  ALT - increase by factor, Any(SCR), GRADE 1 | 6 | 3 | 1 | 6
  ALT - increase by factor, Any(SCR), GRADE 2 | 0 | 0 | 0 | 2
  ALT - increase by factor, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 116 | 120 | 123 | 117
  ALT - increase by factor, Grade 0(SCR), GRADE 0 | 113 | 117 | 122 | 112
  ALT - increase by factor, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 116 | 120 | 123 | 117
  ALT - increase by factor, Grade 0(SCR), GRADE 1 | 3 | 3 | 1 | 4
  ALT - increase by factor, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 116 | 120 | 123 | 117
  ALT - increase by factor, Grade 0(SCR), GRADE 2 | 0 | 0 | 0 | 1
  ALT - increase by factor, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 6 | 4 | 3 | 9
  ALT - increase by factor, Grade 1(SCR), GRADE 0 | 4 | 4 | 3 | 6
  ALT - increase by factor, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 6 | 4 | 3 | 9
  ALT - increase by factor, Grade 1(SCR), GRADE 1 | 2 | 0 | 0 | 2
  ALT - increase by factor, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 6 | 4 | 3 | 9
  ALT - increase by factor, Grade 1(SCR), GRADE 2 | 0 | 0 | 0 | 1
  ALT - increase by factor, Grade 2(SCR), GRADE 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  ALT - increase by factor, Grade 2(SCR), GRADE 1 | 1 | 0 | 0 | 0
  AST - increase by factor, Any(SCR), GRADE 0 | 121 | 122 | 125 | 121
  AST - increase by factor, Any(SCR), GRADE 1 | 2 | 2 | 1 | 3
  AST - increase by factor, Any(SCR), GRADE 2 | 0 | 0 | 0 | 2
  AST - increase by factor, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 120 | 123 | 125 | 122
  AST - increase by factor, Grade 0(SCR), GRADE 0 | 118 | 121 | 125 | 118
  AST - increase by factor, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 120 | 123 | 125 | 122
  AST - increase by factor, Grade 0(SCR), GRADE 1 | 2 | 2 | 0 | 3
  AST - increase by factor, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 120 | 123 | 125 | 122
  AST - increase by factor, Grade 0(SCR), GRADE 2 | 0 | 0 | 0 | 1
  AST - increase by factor, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 3 | 1 | 1 | 4
  AST - increase by factor, Grade 1(SCR), GRADE 0 | 3 | 1 | 0 | 3
  AST - increase by factor, Grade 1(SCR), GRADE 1: number analyzed (Participants) | 3 | 1 | 1 | 4
  AST - increase by factor, Grade 1(SCR), GRADE 1 | 0 | 0 | 1 | 0
  AST - increase by factor, Grade 1(SCR), GRADE 2: number analyzed (Participants) | 3 | 1 | 1 | 4
  AST - increase by factor, Grade 1(SCR), GRADE 2 | 0 | 0 | 0 | 1
  Blood Urea Nitrogen, Any(SCR), GRADE 0 | 123 | 123 | 126 | 125
  Blood Urea Nitrogen, Any(SCR), GRADE 1 | 0 | 0 | 0 | 1
  Blood Urea Nitrogen, Any(SCR), GRADE 2 | 0 | 1 | 0 | 0
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 0: number analyzed (Participants) | 123 | 124 | 125 | 125
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 0 | 123 | 123 | 125 | 124
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 1: number analyzed (Participants) | 123 | 124 | 125 | 125
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 1 | 0 | 0 | 0 | 1
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 2: number analyzed (Participants) | 123 | 124 | 125 | 125
  Blood Urea Nitrogen, Grade 0(SCR), GRADE 2 | 0 | 1 | 0 | 0
  Blood Urea Nitrogen, Grade 1(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Blood Urea Nitrogen, Grade 1(SCR), GRADE 0 | 0 | 0 | 1 | 0
  Blood Urea Nitrogen, Grade 2(SCR), GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 1
  Blood Urea Nitrogen, Grade 2(SCR), GRADE 0 | 0 | 0 | 0 | 1
  Creatinine, Any(SCR), GRADE 0 | 123 | 124 | 126 | 126
  Creatinine, Grade 0(SCR), GRADE 0 | 123 | 124 | 126 | 126

13. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 4
Time Frame: From Day 1 (vaccination) up to Day 91 and up to Day 181
Population: The analysis was performed on the Exposed Set, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 124 | 126 | 126 | 126
Participants
  SAE - Day 91 | 0 | 0 | 1 | 1
  SAE - Day 181 | 0 | 0 | 1 | 2

14. Secondary Outcome: Neutralizing Antibody (Nab) Titers Against RSV Serotype A
Description: Anti RSV-A neutralizing antibody titers are given as geometric mean titers (GMTs) and expressed as Estimated Dose: serum dilution giving a 60% reduction of the signal compared to a control without serum (ED60), calculated on subjects with anti-RSV-A neutralizing antibody titer equal to or above the assay cut-off 18 ED60.
Time Frame: At pre-vaccination at screening (PRE), 7 days post vaccination (Day 8), 30 days post vaccination (Day 31), 60 days post vaccination (Day 61) and 90 days post vaccination (Day 91)
Population: The analysis was performed on the Per-protocol set which included all vaccinated subjects, meeting all protocol requirements and for whom immunogenicity results were available for the specified assay at the corresponding time-point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 123 | 125 | 126 | 126
Titers
  PRE | 851.1 [732.88 to 988.3] | 921.6 [795.52 to 1067.64] | 868.8 [754.18 to 1000.78] | 746.2 [639.96 to 870.02]
  Day 8: number analyzed (Participants) | 120 | 119 | 120 | 123
  Day 8 | 6720.1 [5861.07 to 7705.03] | 9843.6 [8170.69 to 11858.92] | 12638.3 [10883.83 to 14675.63] | 790.8 [665.49 to 939.62]
  Day 31: number analyzed (Participants) | 121 | 121 | 124 | 122
  Day 31 | 5327.6 [4640.84 to 6116.06] | 7323.3 [6236 to 8600.25] | 7943.4 [6942.16 to 9089.07] | 762.9 [638.74 to 911.18]
  Day 61: number analyzed (Participants) | 121 | 121 | 124 | 120
  Day 61 | 5268.4 [4639.84 to 5982.16] | 6783.1 [5782.42 to 7956.92] | 7575.8 [6633.19 to 8652.41] | 875.6 [734.11 to 1044.4]
  Day 91: number analyzed (Participants) | 116 | 119 | 123 | 118
  Day 91 | 4110.7 [3564.87 to 4740.12] | 5186.7 [4357.63 to 6173.57] | 5067.9 [4451.73 to 5769.4] | 840.0 [717.87 to 982.93]

15. Secondary Outcome: Anti-RSVPreF3 Immunoglobulin G (IgG) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in Enzyme Linked Immunosorbent Assay (ELISA) units per millilitre (EL.U/mL), calculated on subjects with anti-RSVPreF3 antibody concentration equal to or above the assay cut-off 25 EL.U/mL.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
Number analyzed (Participants) | 123 | 125 | 126 | 126
EL.U/mL
  PRE | 6753 [6032.53 to 7560.61] | 6447 [5822.74 to 7138.39] | 6738 [5954.89 to 7625.01] | 5583 [5014.96 to 6215.1]
  Day 8: number analyzed (Participants) | 120 | 119 | 120 | 123
  Day 8 | 83187 [75159.55 to 92072.87] | 111915 [97936.91 to 127887.72] | 145984 [131579.66 to 161966.03] | 5902 [5270.51 to 6609.37]
  Day 31: number analyzed (Participants) | 121 | 121 | 124 | 123
  Day 31 | 66153 [58990.44 to 74184.52] | 85096 [75185.08 to 96313.02] | 94360 [86517.06 to 102912.86] | 5856 [5165.49 to 6639.47]
  Day 61: number analyzed (Participants) | 121 | 121 | 124 | 120
  Day 61 | 55170 [49687.49 to 61258] | 65007 [57805.13 to 73106.25] | 71401 [66038.58 to 77198.53] | 6100 [5355.93 to 6948.09]
  Day 91: number analyzed (Participants) | 116 | 119 | 123 | 118
  Day 91 | 39602 [34650.65 to 45261.85] | 47629 [41925.98 to 54108.51] | 51424 [46747.32 to 56569.61] | 6692 [5722.81 to 7825]

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected during the 7-day follow-up period and unsolicited adverse events during the 30-day follow-up period. Serious adverse events were collected from Day 1 up to Day 181.
Arm/Group | RSV MAT Formulation 1 Group | RSV MAT Formulation 2 Group | RSV MAT Formulation 3 Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/126 | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/126 | 1/126 | 2/126
Other Adverse Events (participants affected / at risk) | 94/124 | 96/126 | 105/126 | 83/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV MAT Formulation 1 Group (N=124) | RSV MAT Formulation 2 Group (N=126) | RSV MAT Formulation 3 Group (N=126) | Control Group (N=126)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV MAT Formulation 1 Group (N=124) | RSV MAT Formulation 2 Group (N=126) | RSV MAT Formulation 3 Group (N=126) | Control Group (N=126)
Injection site pain (General disorders) | 59 (59) | 64 (64) | 67 (67) | 20 (20)
Fatigue (General disorders) | 42 (43) | 49 (49) | 41 (41) | 38 (38)
Injection site inflammation (General disorders) | 8 (8) | 14 (14) | 10 (10) | 1 (1)
Injection site swelling (General disorders) | 5 (5) | 7 (7) | 6 (6) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 43 (50) | 53 (57) | 63 (70) | 38 (50)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermohyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 30 (30) | 29 (29) | 23 (23) | 27 (27)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 7 (7) | 10 (11) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 4 (4) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (1)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03674177/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT03674177/SAP_001.pdf